CLINICAL TRIAL: NCT05754138
Title: Safety of Sports for Patients With a Subcutaneous Implantable Cardioverter Defibrillator
Acronym: SPORT-SICD
Status: Recruiting | Type: Observational
Sponsor: Eli Sprecher, MD (Other Government)
Responsible Party: Sponsor-Investigator, Eli Sprecher, MD, Deputy director general for R&D, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: 0132-22-tlv
Record Dates: First submitted 2023-02-11; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Patients With an Implanted S-ICD Who Continue to Exercise Regularly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study population: The study population will consist of patients with an implanted S-ICD as their first implanted device, who continue to exercise regularly and actively participate in competitive or recreational sports with a sport-intensity above a predefined level
  Interventions: Device: Sport SICD

INTERVENTIONS:
Device: Sport SICD — Follow up

SUMMARY:
A multicenter observational study designed specifically to collect data on the safety of sport activities in patients with implanted S-ICD systems.

DETAILED DESCRIPTION:
Observational multicenter study with prospective follow-up but accepting also retrospectively collected data. Data will be collected and entered in a secure dedicated web-based database.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (male or female) is <60 years of age.
2. Patient has an implanted with a new-generation S-ICD [Boston Scientific EMBLEM, Generations 2 (model A209), 3 (A219) or newer].
3. Present device is the first defibrillator implanted.
4. Patient has a functioning LATITUDE™ Home-Monitoring-System at home, knows how to use it and sends weekly reports via the home-monitoring system.
5. Patient actively participates in sport activities above a predefined level of exercise (see below).
6. Patient understands that, at present, there is virtually no data on the safety of sport participation for patients with implanted S-ICD system, particularly regarding potential damage caused by sport activities to the S-ICD system, including the subcutaneous electrode.
7. Patient understands that the level of sport activity, type of sport and frequency of exercise activities are entirely at his/her own discretion and responsibility.
8. Patient understands that The Sport S-ICD Study investigator neither encourage nor discourage performance of any given sport.
9. Patient understands that The Sport S-ICD Study is not liable for- and does assume any responsibility for any damages caused by sport participation to the implanted system or the health of patients participating in the study.
10. Patient is willing to provide informed consent to participate in the SPORT S-ICD Study. Informed consent includes agreement to provide all the following information:

    1. Clinical data (age, gender, clinical diagnosis, indication for S-ICD implantation, arrhythmic events since S-ICD implantation, adverse events since S-ICD implantation)
    2. Type and level of exercise and sport participation at the time of inclusion and during follow-up.
    3. Information concerning endpoint events during follow-up.
    4. Direct access to the patients' LATITUDE™ Home-Monitoring-System data, both at the time of inclusion and all weekly reports during the follow-up period, until the study ends or the informed consent is revoked. Access to the personal LATITUDE™ Home-Monitoring-System data is in addition to the access by the primary treating physician and only for purpose of data collection for the study. Consent from the patient AND for the primary treating physician (monitoring the patient's LATITUDE data) are required. Once the study ends, participating patients will be notified that the Study Investigators are no longer monitoring his/her LATITUDE Home-Monitoring-System.

Exclusion Criteria:

1. Subjects with an inability to communicate well with the investigators.
2. Subjects who are non-cooperative or unwilling to sign consent form.
3. Evidence suggestive of malfunction of the implanted S-ICD system (like abnormal impedance or detected noise) at the time of screening

Ages: 10 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: patients with an implanted S-ICD as their first implanted device, who continue to exercise regularly and actively participate in competitive or recreational sports with a sport-intensity above a predefined level
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Tachyarrhythmia-related death or externally resuscitated cardiac arrest due to S-ICD | 5 years
  Quantitative data will be reported by S-ICD interrogation including shock failure, incessant ventricular arrhythmia, or post-shock pulseless electrical activity.

SECONDARY OUTCOMES:
S-ICD Lead fracture/malfunction | 5 years
  Noise/impedance will be reported by S-ICD interrogation

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No